CLINICAL TRIAL: NCT07172217
Title: Clinical Study on the Efficacy and Safety of Disitamab Vedotin Combined With Iparomlimab and Tuvonralimab in the Second-Line Treatment of HER2-Expressing Recurrent Cervical Cancer
Brief Title: The Efficacy and Safety RC48 Plus QL1706 in Second-Line Treatment of HER2-Expressing Recurrent CC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Li Peng, Department of Gynecology, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202503-017-1
Record Dates: First submitted 2025-08-28; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Cervical Cancer
Keywords: RC48;QL1706;HER2-Expressing;Recidivation; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 and QL1706 (Experimental)
  Interventions: Drug: RC48; Drug: QL1706

INTERVENTIONS:
Drug: RC48 — Disitamab Vedotin (RC48) : 2.5 mg/kg, administered once every 3 weeks (Q3w), via intravenous infusion on Day 1 of each treatment cycle
Drug: QL1706 — Drug: QL1706 Iparomlimab and Tuvonralimab (QL1706) : 5 mg/kg in total, administered once every 3 weeks (Q3w), via intravenous infusion on Day 1 of each treatment cycle

SUMMARY:
This is a single-arm study. The efficacy and safety of Disitamab Vedotin combined with Apalutamide and Toripalimab in the second-line treatment of HER2-expressing recurrent cervical cancer are evaluated based on the following indicators:

Primary evaluation indicator: Objective Response Rate (ORR)

Secondary evaluation indicators:

Efficacy-related indicators: Progression-Free Survival (PFS), Disease Control Rate (DCR), Duration of Response (DOR), Overall Survival (including median Overall Survival [mOS] and 1-year, 2-year, 3-year Overall Survival rates) Safety-related indicators: Adverse Events (AEs) and Serious Adverse Events (SAEs).

DETAILED DESCRIPTION:
This study is a multicenter, open-label, single-arm, exploratory trial. It enrolls 33 participants with recurrent cervical cancer who have HER2 expression (IHC 1+, 2+, or 3+). After eligible participants are enrolled, they will receive treatment with RC48 (dose: 2.5mg/kg, Q3W, intravenous infusion) in combination with QL1706 (dose: 5mg/kg, Q3W, intravenous infusion), with a treatment window of ±3 days. During the study, safety assessment and efficacy assessment will be conducted.

Safety Assessment For participants who have received at least one dose of the study drug, the safety assessment will start from the administration of the study drug. It will be performed before each drug administration, assessed once every 3 weeks (with a window of ±3 days), and continue until 30 days after the last dose of the study drug or the initiation of new anti-tumor treatment.

Efficacy Assessment Tumor assessment will be conducted in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Starting from the administration of the study drug, assessments will be performed once every 6 weeks (with a window of ±3 days) until the occurrence of intolerable toxicity or radiologically confirmed disease progression.

For participants who experience disease progression or start other anti-tumor treatments, survival follow-up will be conducted once every 3 months (with a window of ±14 days) from the date of confirmation. Information on the participants' subsequent anti-tumor treatment and survival status will be collected until the participant's death, withdrawal of informed consent, loss to follow-up, study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily enroll in the study and sign a written informed consent form;
* Female patients aged 18 to 75 years (inclusive);
* Histologically or cytologically confirmed primary cervical squamous cell carcinoma, adenocarcinoma, adenosquamous carcinoma, or small cell (neuroendocrine) cervical cancer;
* Progressive disease or recurrent disease after first-line treatment for recurrent cervical cancer;
* Subjects can provide tumor specimens (paraffin blocks, formalin-fixed paraffin-embedded [FFPE] sections, or fresh tissue sections) from the primary or metastatic site for HER2 detection, with HER2 immunohistochemistry (IHC) test results of IHC 1+, 2+, or 3+ (previous test results confirmed by the investigator are also acceptable);
* Presence of at least one evaluable lesion (per RECIST 1.1 criteria);
* Expected survival time ≥ 6 months;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 1;
* For female patients of childbearing potential (i.e., premenopausal or not surgically sterilized), the serum pregnancy test result within 7 days before the first administration of the study drug must be negative; and reliable contraceptive measures must be used during the study drug administration period and within 60 days after the last dose;
* Normal function of major organs, meeting the following criteria:

Left ventricular ejection fraction (LVEF) ≥ 50%; Hemoglobin (Hb) ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelets (PLT) ≥ 100 × 10⁹/L; Serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN in the absence of liver metastasis, and ALT and AST ≤ 5 × ULN in the presence of liver metastasis; Serum creatinine (Scr) ≤ 1.5 × ULN, or creatinine clearance (CrCl) ≥ 40 mL/min calculated by the Cockcroft-Gault formula.

Exclusion Criteria:

* History of malignant tumors other than cervical cancer, except for the following two situations:

  1. Patients who have received potentially curative treatment and have no evidence of the disease for 5 years;
  2. Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, cervical carcinoma in situ, and other carcinoma in situ that have been successfully treated with resection;
* Previous allogeneic stem cell or solid organ transplantation;
* Previous systemic anti-tumor therapy (including traditional Chinese medicine with anti-tumor indications) completed less than 4 weeks before the first administration of the study drug, or patients whose adverse events caused by previous treatment have not recovered to ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) (except for alopecia and pigmentation);
* Vaccination with live vaccines within 4 weeks before the start of study drug administration, or planned receipt of any vaccines (except COVID-19 vaccines) during the study period;
* Previous or current history of congenital or acquired immunodeficiency diseases;
* Previous treatment with other antibody-drug conjugates (ADCs);
* Patients with known or suspected history of allergy to recombinant humanized anti-HER2 monoclonal antibody-MMAE conjugates and anti-PD-1 drugs of the same class, or history of hypersensitivity to chimeric/humanized antibodies or fusion proteins, or allergy to the excipients of the study drug;
* Other significant clinical and laboratory abnormalities that the investigator deems may affect safety evaluation, such as uncontrolled diabetes mellitus, chronic kidney disease, peripheral neuropathy of Grade 2 or higher (per CTCAE V5.0), abnormal thyroid function, etc.;
* Heart failure of New York Heart Association (NYHA) Class 3 or higher;
* Severe infection in active stage or with poor clinical control; active infections include:

  1. Positive for human immunodeficiency virus (HIV) (HIV1/2 antibodies);
  2. Active hepatitis B (positive for hepatitis B surface antigen [HBsAg], or hepatitis B virus deoxyribonucleic acid [HBV DNA] > 2000 IU/ml with abnormal liver function);
  3. Active hepatitis C (positive for hepatitis C virus [HCV] antibodies, or HCV ribonucleic acid [HCV RNA] ≥ 10³ copies/ml with abnormal liver function);
  4. Active tuberculosis;
  5. Other uncontrolled active infections (Grade > 2 per CTCAE V5.0); Unrecovered from surgery (e.g., presence of unhealed surgical incisions or severe postoperative complications);
* Other circumstances deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 months after the last subject participating in
  The proportion of subjects with complete response (CR) and partial response (PR) according RESIST 1.1 in total subjects.

SECONDARY OUTCOMES:
Progression-Free Survival | Approximately 1 years after last participant enrollment.
  The time elapsed from the enrollment date to the first occurrence of either tumor progression or death from any cause.
disease control rate (DCR) | Approximately 1 years after last participant enrollment.
  The proportion of subjects with complete response (CR) and partial response (PR) and stable disease(SD) in total subjects
duration of response (DOR) | The time from the start of treatment to the first observation of response (Complete Response [CR] or Partial Response [PR]) that is ultimately confirmed (typically via a subsequent reassessment at least 4 weeks later, per RECIST criteria).
  The time from the date for first documented response of complete response (CR) or partial response (PR) to the date of first documented of disease progression or death, whichever occurs first.
overall survival (OS) | Approximately 1 years after last participant enrollment.
  The time from the starting date of study drug to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Ji'an, Shandong, China

IPD SHARING:
Plan to Share IPD: No